CLINICAL TRIAL: NCT05628987
Title: The Association of Gut Microbiota and Spermatogenic Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Hongwei Zhou, Professor, Zhujiang Hospital
Other Study IDs: Zhujiangjj-03
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Infertility, Male; Azoospermia; Oligozoospermia; Asthenozoospermia; Teratozoospermia
Keywords: Microbiota; Infertility, Male; Sperm
MeSH Terms: conditions — Infertility, Male; Azoospermia; Oligospermia; Asthenozoospermia; Teratozoospermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Feces, urine, blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Azoospermia: After an abstinence period of 2-7 days, two basic semen analysis, the absence of spermatozoa
  Interventions: Other: no intervention
- Oligozoospermia: After an abstinence period of 2-7 days, the total sperm number <39*10^6 per ejaculate or the sperm concentration < 15 * 10^6 per ml
  Interventions: Other: no intervention
- Asthenozoospermia: After an abstinence period of 2-7 days, the progressive motility (PR) < 32%
  Interventions: Other: no intervention
- Teratozoospermia: After an abstinence period of 2-7 days, the percentage of morphologically normal spermatozoa <4%
  Interventions: Other: no intervention
- Control: After an abstinence period of 2-7 days, the basic semen analysis is normal.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Observational studies, no intervention

SUMMARY:
This is a multicenter, case-control study that aims to investigate the relationship between microbiota and sperm quality via stool, blood, and urine microbiome, metabolomics, and collected clinical metadata. The results of the spermatogenic dysfunction, including aspermia, oligozoospermia, asthenozoospermia, and teratozoospermia, will be compared to normal basic semen analysis utilizing the World Health Organization (WHO) semen analysis procedure 5th edition.

DETAILED DESCRIPTION:
Infertility is a global issue that affects as much as 10%-15% of couples. Approximately half of infertility can be attributed to men. Recently, a worldwide accelerated decline in sperm counts was reported. And the gut microbiome modulates many physiological functions and diseases, including host immunity, metabolic diseases, neuropsychiatric disorders, and so on. Recent publications demonstrate the links between intestinal microbiota and sperm production in fat animals and a few patients. And systemic clinical research would be necessary to explore the human microbiota and males with fertility disorders.

The primary objective of the study is to determine the links between the gut microbiome and sperm quality utilizing microbiome and metabolomics. Stool, blood, and urine will be collected when a patient completes basic semen analysis and informed consent is signed. Microbiome and metabolomics will be compared among aspermia, oligozoospermia, asthenozoospermia, teratozoospermia, and normal individuals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years, males
* Body Mass Index (BMI):18.5-29.9 kg/m^2
* After an abstinence period of 2-7 days, two abnormal semen analysis, the absence of spermatozoa from both replicates will be included in the azoospermia group, the total sperm number (<39*10^6 per ejaculate) or the sperm concentration ( < 15 * 10^6 per ml) will be oligozoospermia group, the progressive motility (PR) (< 32%) will be asthenozoospermia group; the percentage of morphologically normal spermatozoa (<4%) will be teratozoospermia group
* Willing to provide feces, urine, blood samples, able to complete study questionnaires aimed at lifestyle factors (cigarette smoking, high temperature environment and others ) and other data collection instruments (e.g. physical activity, food frequency questionnaire, stress and others)

Exclusion Criteria:

* Age < 18 or > 45 years
* History of Zocanidin, Vitamin E, antibiotics, clyster, gastrointestinal endoscope in the past 30 days, or other drugs known to interact with semen quality or gut microbiota, history of high alcohol consumption (liquor over 200 ml, beer over 1000 ml) in the past 7 days or drinking every week in the past month
* A known genetic cause of male factor spermatogenesis dysfunction, including chromosomal or gene disorders (e.g. Y chromosome deletions, CFTR mutation)
* History of male reproductive system (e.g. testis, epididymis, seminiferous duct and others) damage, surgery, tumor or infection
* History of Crohn's disease, ulcerative colitis, acute gastrointestinal disease, renal failure, liver cirrhosis, hypoplasia, X-rays exposure and other diseases related to spermatogenic dysfunction, history of intestinal gastrointestinal surgery (exclude appendix surgery)
* History of psychoses or other mental conditions that would result in cognitive impairment and inability to participate in any part of this study including the informed consent process

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers and patients will be recruited from the outpatient clinics of the Department of Andrology, Reproduction in our participant hospitals. Patients are from licensed doctor of the clinical research center. The age of healthy volunteers and patients in the same hospital will be matched.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Microbiome | Baseline
  The microbial composition of the stool samples was determined by 16S rRNA (ribosomal ribonucleic acid) gene sequencing analysis and metagenomics. Comparison of microbial abundance and diversity of healthy volunteers and patients with spermatogenic dysfunction.
Metabolomics | Baseline
  Metabolomics is the large-scale study of small molecules, such as fatty acids, bile acids, lipid mediators and others. Comparison of metabolites of healthy volunteers and patients with spermatogenic dysfunction.

SECONDARY OUTCOMES:
Physical activity time | Baseline
  Analyzing physical activity (hours/week) of different groups. The questionnaire about Physical Activity Time, "Over the past 30 days, on average how many hours per week did you usually spend on physical activity?"
Daily sitting time | Baseline
  Analyzing daily sitting time (hours) of different groups. The questionnaire about Daily Sitting Time, "Over the past 7 days, on average how many hours did you usually spend sitting on a typical day?"
Eating habits | Baseline
  Analyzing eating habits (vegetarian or meat lover) of different groups.
Sleeping time | Baseline
  Analyzing daily sleeping time (hours) of different groups. The questionnaire about Sleeping Time, "Over the past 7 days, on average how many hours did you usually sleep per day?"
Education level | Baseline
  Analyzing education level (highest grade or level of school) of different groups. The questionnaire about Education Level, "What is the highest grade or level of school you have completed or the highest degree you have received? The response categories are: less than 9th grade education, 10-12th grade education (includes no diploma), some college or associates (AA) degree, and college graduate or higher."
Family income (CNY) | Baseline
  Analyzing annual family income (CNY) of different groups. The questionnaire about Family Income, "How much is annual family income (CNY)?"
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  Analyzing Patient Health Questionnaire-9 (PHQ-9) scores of different groups. The Patient Health Questionnaire 9 (PHQ-9) is one of the tools used to screen for the presence and severity of depression. Each response category of 'not at all', 'several days', 'more than half the days' and 'nearly every day' is assigned a score of 0, 1, 2 and 3 respectively. The total score is calculated by adding together the scores for the 9 questions. The final scores of 0-4, 5-9, 10-14, 15-19, 20-27 are the ranges for none, mild, moderate, moderately severe and severe, respectively.
Years of smoking | Baseline
  Analyzing years of smoking of different groups. The questionnaire about Years of Smoking, "For about how many years have you smoked? 0 means non-smoker"
Number of cigarettes smoked | Baseline
  Analyzing number of cigarettes smoked of different groups. The questionnaire about Number of Cigarettes Smoked, "During the past 30 days, on average how many cigarettes did you smoke per day? non-smoker choose 0"
History of drinking in the past one month | Baseline
  Analyzing history of drinking of different groups in the past one month. "Considering all types of alcoholic beverages, during the past one month, do you have at least 1 drink of any kind of alcohol per week, not counting small tastes or sips? By a drink, I mean 500 ml beer, 50 ml liquor, or 500ml other type of alcoholic beverage."
History of drinking in the past 7 days | Baseline
  Analyzing history of drinking of different groups in the past 7 days. "Considering all types of alcoholic beverages, during the past 4 weeks, do you have at least 1 drink of any kind of alcohol, not counting small tastes or sips? By a drink, I mean 1000 ml beer, 200 ml liquor, or 1000ml other type of alcoholic beverage.""Considering all types of alcoholic beverages, during the past one month, do you have at least 1 drink of any kind of alcohol per week, not counting small tastes or sips? By a drink, I mean 500 ml beer, 50 ml liquor, or 500ml other type of alcoholic beverage."
Body Mass Index (BMI) | Baseline
  To analyze Body Mass Index (kg/m^2) of different groups, height(cm) and weight(kg) will be measured.
Waistline | Baseline
  Analyzing waistline (cm) of different groups.
Spermatic concentration | Baseline
  To analyze spermatic concentration (10^6 per ml). According to the World Health Organization (WHO) semen analysis procedure 5th edition, spermatic concentration will be measured.
Total sperm count | Baseline
  To analyze total sperm count (10^6 per ejaculate). According to the World Health Organization (WHO) semen analysis procedure 5th edition, total sperm count will be measured.
Spermatic progressive motility | Baseline
  To analyze spermatic progressive motility (%). According to the World Health Organization (WHO) semen analysis procedure 5th edition, progressive motility will be measured.
Percentage of normal morphology of sperm | Baseline
  To analyze percentage of normal morphology of sperm (%). According to the World Health Organization (WHO) semen analysis procedure 5th edition, percentage of normal morphology of sperm will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Study Chair — Southern Medical University, China
Locations (3):
- China (3):
  - Guangdong Provincial Fertility Hospital, Guangzhou, Guangdong
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He Y, Wu W, Zheng HM, Li P, McDonald D, Sheng HF, Chen MX, Chen ZH, Ji GY, Zheng ZD, Mujagond P, Chen XJ, Rong ZH, Chen P, Lyu LY, Wang X, Wu CB, Yu N, Xu YJ, Yin J, Raes J, Knight R, Ma WJ, Zhou HW. Regional variation limits applications of healthy gut microbiome reference ranges and disease models. Nat Med. 2018 Oct;24(10):1532-1535. doi: 10.1038/s41591-018-0164-x. Epub 2018 Aug 27. PMID 30150716
- [Background] Yang H, Zhang J, Xue Z, Zhao C, Lei L, Wen Y, Dong Y, Yang J, Zhang L. Potential Pathogenic Bacteria in Seminal Microbiota of Patients with Different Types of Dysspermatism. Sci Rep. 2020 Apr 23;10(1):6876. doi: 10.1038/s41598-020-63787-x. PMID 32327694
- [Background] Ding N, Zhang X, Zhang XD, Jing J, Liu SS, Mu YP, Peng LL, Yan YJ, Xiao GM, Bi XY, Chen H, Li FH, Yao B, Zhao AZ. Impairment of spermatogenesis and sperm motility by the high-fat diet-induced dysbiosis of gut microbes. Gut. 2020 Sep;69(9):1608-1619. doi: 10.1136/gutjnl-2019-319127. Epub 2020 Jan 2. PMID 31900292
- [Background] Martinot E, Thirouard L, Holota H, Monrose M, Garcia M, Beaudoin C, Volle DH. Intestinal microbiota defines the GUT-TESTIS axis. Gut. 2022 Apr;71(4):844-845. doi: 10.1136/gutjnl-2021-324690. Epub 2021 May 13. No abstract available. PMID 33985968